CLINICAL TRIAL: NCT04153474
Title: Exit Strategy After Percutaneous Nephrolithotomy: Large or Small Bore Tube? Randomised Controlled Trial
Brief Title: Exit Strategy After Percutaneous Nephrolithotomy: Large or Small Bore Tube?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Shoma, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP-LP PCNL
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-10

CONDITIONS: Urolithiasis; Nephrolithotomy; Percutaneous Nephrolithotomy (PNL); Nephrostomy Tube (NT); Pain
Keywords: Percutaneous nephrolithotomy (PNL); Nephrostomy tube (NT); Pain; Patient satisfaction
MeSH Terms: conditions — Urolithiasis; Pain; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- large-bore nephrostomy tube (LBNT) (Active Comparator): large-bore 22 french nephrostomy tube (LBNT)
  Interventions: Procedure: large-bore nephrostomy tube (LBNT)
- small-bore nephrostomy tube (SBNT) (Active Comparator): small-bore 14 french nephrostomy tube (SBNT)
  Interventions: Procedure: small-bore nephrostomy tube (SBNT)

INTERVENTIONS:
Procedure: large-bore nephrostomy tube (LBNT) — large-bore 22 french nephrostomy tube (LBNT)
  Other Names: LBNT
  Arms: large-bore nephrostomy tube (LBNT)
Procedure: small-bore nephrostomy tube (SBNT) — small-bore 14 french nephrostomy tube (SBNT)
  Other Names: SBNT
  Arms: small-bore nephrostomy tube (SBNT)

SUMMARY:
Regarding to the distribution of nephrostomy tube (NT) size usage by country. There was a clear distinction between countries that used solely the small bore (SB) NT (Chile and Australia) and those that used solely the large bore (LB) NT (Czech Republic and Japan). There is also a trend toward SB NT in North America (~75% in USA and Canada) and toward LB NT in South America (~80% in Argentina and Mexico). In Europe the trend is equal (~50% in Germany, France, Greece and UK). Based on previous data and in view of conflicting data about postoperative complication including extravasation, bleeding and hemoglobin change and pain between previous studies, we will conduct this randomised trial comparing SB and LB NT following PNL.

Our aim to evaluate the safety of small versus large bore NT reporting complications using the Clavien-Dindo system with categorisation of PNL-specific complications

ELIGIBILITY:
Inclusion Criteria:

1. Staghorn calculi
2. Renal pelvis stones =>2 cm
3. Lower pole stones= >1.5 cm
4. upper ureteral calculi =>1.5 cm
5. SWL-resistant stones

Exclusion Criteria:

1. Age <18 years or Pregnancy
2. Tubeless PNL
3. Need for 3 percutaneous tracts intraoperative
4. Morbid obesity (BMI >40)
5. Refuse to complete study requirements
6. Tumour in the presumptive access tract area or Potential malignant kidney tumour

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of hemoglobin reduction difference between groups | 8 months
  measured in gram/liter

SECONDARY OUTCOMES:
postoperative pain score | 8 months
  Assessed by Visual Analogue Scale (VAS) points from 0 to 10
postoperative patient satisfaction | 8 months
  measured by The Freiburg Index of Patient Satisfaction (FIPS score) from 1 to 6
overall postoperative complication | 8 months
  assesed by Clavien-Dindo system

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: No